CLINICAL TRIAL: NCT01333332
Title: Phase II Trial of Accelerated Fraction Radiotherapy With Concomitant Capecitabine as Neoadjuvant Therapy of Resectable and Borderline Resectable Pancreas Cancer
Brief Title: Radiotherapy With Chemotherapy as Neoadjuvant Therapy of Resectable and Borderline Resectable Pancreas Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Hanna K. Sanoff, MD, Assistant Professor, Principal Investigator, University of Virginia, Department of Medicine, Hematology and Oncology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15050
Record Dates: First submitted 2011-03-04; First posted 2011-04-11 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2011-04

CONDITIONS: Pancreatic Cancer
Keywords: Pancreas; Radiation
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Capecitabine, Radiation (Experimental)
  Interventions: Drug: Capecitabine; Radiation: Standard Dose Acclerated Fraction Radiotherapy

INTERVENTIONS:
Drug: Capecitabine — Capecitabine
Radiation: Standard Dose Acclerated Fraction Radiotherapy — Standard dose accelerated fraction radiotherapy

SUMMARY:
The purpose of this study is to determine safety and to obtain preliminary estimates of the rate of major pathologic response of neoadjuvant accelerated fraction, standard dose radiation given with chemotherapy in patients with locally advanced pancreas cancer.

ELIGIBILITY:
Inclusion:

1. Clinically staged I-III, pathologically confirmed adenocarcinoma of the pancreas. Mixed (e.g. adeno-squamous, neuroendocrine features) and/or poorly differentiated carcinomas are eligible as long as the carcinoma is not a predominantly neuroendocrine carcinoma. Cancers must be deemed by multidisciplinary assessment at UVA to be either

   * Resectable

     * No overt evidence of vascular involvement
     * No overt metastatic disease
   * Borderline Resectable, meeting one of the following categories:

     * Local tumor characteristics:

       * Abutment of <180◦ of the superior mesenteric artery and/or celiac axis
       * Abutment or encasement of a short segment hepatic artery
       * Involvement of the portal vein or superior mesenteric vein amenable to vascular reconstruction
     * Concern for extra pancreatic metastatic disease

       * indeterminant nodule on imaging
       * Pathologically confirmed N1
     * Borderline performance status or medical comorbidities as determined by investigators to be concerning for patient's ability to tolerate pancreatic resection
   * Patients with overtly unresectable disease are ineligible
2. No prior therapy for pancreatic cancer, including surgery, radiation, or chemotherapy
3. ≥18 years of age
4. Able to provide informed consent and comply with study procedures
5. Concurrent therapy with warfarin is permitted, but INR must be checked weekly
6. Concurrent therapy with phenytoin is permitted, but phenytoin levels must be checked weekly.
7. Concurrent therapy with CYP2C9 substrates is permitted but discouraged. Patients taking fluoxetine, glipizide, losartan, voriconazole, or other CYP2C9 substrates should consider switching to an alternative medication if feasible. (see Appendix 11.3 for a list of CYP2C9 substrates).
8. Adequate organ function:

   * Hematologic

     * ANC ≥ 1.5 x 10^9 cells/liter
     * Plts ≥ 100,000 x 10^9 cells/liter
   * Hepatic

     * Total bilirubin ≤ 5 fold the upper limits of normal for laboratory if due to biliary obstruction secondary to disease. For patients with total bilirubin 3-5 times the upper limit, attempt to relieve biliary obstruction is required
     * AST/ALT ≤ 5 fold the upper limits of normal for laboratory
   * Renal

     * Creatinine clearance as measured by Cockcroft-Gault (APPENDIX) of >30 mL/min.
     * Patients with creatinine clearance of 30-50 mL/min require 25% reduction of capecitabine dose.

Exclusion:

1. No pregnant or lactating women. Women of child bearing age must have a negative pregnancy test within seven days of beginning therapy and agree to use reliable contraception for the duration of the study period.
2. No comorbid condition which is deemed by the investigator to have a life expectancy of less than 6 months
3. No other malignancy diagnosed within the past 5 years, excepting all in situ cancers and invasive nonmelanomatous skin cancers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2010-08; Primary Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
To determine the safety of neoadjuvant accelerated fraction standard dose radiotherapy to 50 Gy with concomitant capecitabine in patients with resectable and borderline resectable pancreas cancer. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States